CLINICAL TRIAL: NCT01538147
Title: Association Between Restless Leg Syndrome and Severe Preeclampsia. A Case Control Study.
Brief Title: Restless Leg Syndrome and Severe Preeclampsia
Status: Completed | Type: Observational
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., MD, Saint Thomas Hospital, Panama
Other Study IDs: MHST2012-02
Record Dates: First submitted 2012-02-19; First posted 2012-02-23 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Restless Leg Syndrome; Severe Preeclampsia
Keywords: Restless Leg Syndrome; Severe Preeclampsia
MeSH Terms: conditions — Restless Legs Syndrome; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with Severe preeclampsia
- Control: Patients with normal pregnancies at term

SUMMARY:
Restless Leg Syndrome is a common but not well recognized central nervous system disorder. It is more prevalent during pregnancy and, if present before pregnancy, can develop an exacerbation of symptoms. In some of the hypothesis trying to explain this syndrome, the physiopathology can also explain hypertensive disorders of pregnancy. So far, no study has been done trying to link both disorders.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24-34 weeks
* Severe preeclampsia

Exclusion Criteria:

* Neurological disorders (central nervous system)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients with severe preeclampsia (cases) and normal pregnancies at term (control).
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Restless Leg Syndrome | 10 months
  Number of patients with criteris for the diagnosis of Restless Leg Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo A Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama